CLINICAL TRIAL: NCT06112483
Title: SWELE Programme: An Unstructured Outdoor Play With Mindfulness-based Interventions to Promote Mental Health Among Children and Adolescents With Special Education Needs
Brief Title: SWELE Program: An Unstructured Outdoor Play With Mindfulness-based Interventions to Promote Mental Health Among Students With Special Education Needs
Acronym: SEN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, LEE Regina Lai Tong, Professor, Chinese University of Hong Kong
Other Study IDs: 2022.659-T
Record Dates: First submitted 2023-08-21; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Specific Learning Disorder; Intellectual Disability, Mild to Moderate; Autism Spectrum Disorder; Attention Deficit Hyperactivity Disorder; Physical Disability
Keywords: Unstructured play; Mindfulness-based interventions; Special education needs; Children and adolescents; Emotional; Anxiety; Depression; Self-regulation
MeSH Terms: conditions — Specific Learning Disorder; Intellectual Disability; Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Anxiety Disorders; Depression; Self-Control

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and adolescents with special education needs: Children and adolescents with special education needs, including (a) specific learning difficulties; (b) intellectual disability; (c) autism; (d) attention deficit hyperactivity disorder; (e) physical disabilities.
  Interventions: Behavioral: SWELE Programme

INTERVENTIONS:
Behavioral: SWELE Programme — This 16-week programme focuses on Supporting Wellness in E-Child Learning Environments (SWELE) programme by combining unstructured outdoor play with mindfulness-based interventions to promote mental health in SEN students, in the context of the COVID-19 pandemic. There is no such SWELE programme to promote mental health for SEN students in Hong Kong, especially in the context of COVID-19 pandemic.
  A playful approach of unstructured play has also been found effective on promoting positive emotions and emotional competence among early adolescents (Harn & Bo, 2019). Unstructured Outdoor Play coupled with Mindfulness-based Interventions via SWELE programme to Promote Mental Health for children and adolescents with SEN during COVID-19 pandemic. Very limited unstructured outdoor play-based programme integrated into the extra-curricular activities in the special schools in Hong Kong.
  Other Names: Unstructured play with mindfulness-based interventions

SUMMARY:
This is an observational study with the aim of SWELE Programme is to raise mental health knowledge and awareness by implementing a play-based approach on Supporting Wellness in E-Child Learning Environments (SWELE) programme combining unstructured outdoor play activities with mindfulness-based interventions to promote mental health in children and adolescents with special education needs (SEN), in the context of the COVID-19 pandemic.

This is a 16-week SWELE programme and it will be conducted in two batches. Each batch has three special schools. The main activities include: One training workshop for three groups in each special school: 1) Scout Leaders (special schools' teachers), 2) SEN students (scouts in the school) to become Youth Mental Health Ambassadors and 3) for parents, school social workers, school nurses, schoolteachers and stakeholders; 30 minutes unstructured outdoor play with mindfulness activities 2 times per week for 16 weeks

After participated the SWELE programme, the primary outcomes include reducing anxiety symptoms, reducing negative emotions, improving social skills in peer relationships; and changing in playfulness level among SEN children and adolescents.

Main activities of SWELE programme:

* Unstructured outdoor free play integrated into the school's extra-curricular activities (Youth Mental Health Ambassadors) to promote SEN students' mental health for objectives 1-4.
* Use mindfulness-based podcasts, mindfulness games, mindfulness art for objectives 1-2.
* Through meditation and deep breathing technique, storytelling with relaxing waves piano music, yoga and mindful art for objectives 1-2.
* Training Workshops (Training of trainers) for Scout Leaders who will implement SWELE program in each special school.
* Youth Mental Health Ambassador Program for SEN students who are enrolled in Scout Club in each special school; SWELE training workshops for parents and schoolteachers will also be held in each special school for objectives 1-4.
* Examples of unstructured play might be creative play alone or with others, including artistic or musical games. imaginative games - for example, making cubbyhouses with boxes or blankets, dressing up or playing make-believe, exploring new or favorite spaces like school backyards, parks, playgrounds and so on.

DETAILED DESCRIPTION:
Intervention: SWELE Program:

How does this SWELE programme combine unstructured outdoor play with mindfulness-based interventions is different from other existing services in the community? This 16-week programme focuses on Supporting Wellness in E-Child Learning Environments (SWELE) programme by combining unstructured outdoor play with mindfulness-based interventions to promote mental health in SEN students, in the context of the COVID-19 pandemic. There is no such SWELE programme to promote mental health for SEN students in Hong Kong, especially in the context of COVID-19 pandemic. Six special schools have been recruited and they would participate the SWELE programme.

A playful approach of unstructured play has also been found effective on promoting positive emotions and emotional competence among early adolescents. Unstructured Outdoor Play coupled with Mindfulness-based Interventions via SWELE programme to Promote Mental Health for children and adolescents with SEN during COVID-19 pandemic. Very limited unstructured outdoor play-based programme integrated into the extra-curricular activities in the special schools in Hong Kong.

The COVID-19 pandemic has resulted in increased anxiety and stress among children and adolescents in Hong Kong. In order to help alleviate these symptoms, the project team of the SWELE program is collaborating with The Scout Association of Hong Kong on a 16-week SWELE programme to promote SEN students' mental health. The mindfulness-based interventions focus on social-emotional learning activities in schools. Without intentional social-emotional development, SEN students may not learn how to process their emotions and connect with other in healthy ways. That is where mindfulness can come in. What is mindfulness? Mindfulness involves both an awareness and an acceptance of both the world around us and our internal experiences. Mindful people tend to focus more on the present instead of reflecting on the past or future, and they cultivate a curiosity towards their thoughts, emotions, or physical sensations.

The new knowledge generates from the findings of this mental health promotion project are important for raising the public's awareness about the impact on SEN student's mental health and advancing our understanding of the COVID-19 pandemic's impacts on service disruption and transition and subsequently on concerning SEN students' mental health. Thus, school health policy and strategies should be developed appropriately in promoting SEN

ELIGIBILITY:
Inclusion Criteria

SEN students:

1. are studying in a special school;
2. can speak and understand Cantonese
3. have no diagnosis of any cardiovascular disease
4. can provide parental consent

Exclusion Criteria

SEN students:

1. are not studying in a special school;
2. do not speak and understand Cantonese
3. have been diagnosed with cardiovascular disease
4. do not provide parental consent

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents aged 6-18 years old with mild to moderate physical and intellectual disabilities (SEN students) from six selected special schools. They will be recruited and participated the SWELE Programme.
Sampling Method: Non-Probability Sample
Enrollment: 1064 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-07-14 (Estimated)

PRIMARY OUTCOMES:
Change scores from baseline to 16 weeks in SEN students' mood using the Mood Scale | 16 weeks
  To reduce over 80% of SEN students' low mood after participated the 16-week SWELE programme.
  The Mood Scale includes five different emoji with a 5-points response scale of mood ranging from 1-5: 1-Very bad; 2-bad, 3-so-so, 4-good; to 5-very good. The range of scale score can be from 1 to 5 where higher scores represented very good mood and emotion.
Change scores from baseline to 16 weeks in SEN students' anxiety symptoms using the Chinese version of the short-form State-Trait Anxiety Inventory (STAI-S-6 & STAI-T-7) | 16 weeks
  To reduce over 80% of SEN students' anxiety symptoms after participated the 16-week SWELE programme.
  The Chinese version of short-form of State-Trait Anxiety Inventory (STAI-S-6 & STAI-T-7) demonstrates sound psychometric properties to evaluate the anxiety level. Observers will be asked to rate each item using the following scale (Scale of 1-4; 1 = not at all, 2 = a little, 3 = moderate, 4 = extremely). The range of score from 13 to 52. The mean of the Inventory will be calculated and the mean difference will be compared between the baseline and at 16 weeks. The higher score shows a higher level of anxiety.
Change scores from baseline to 16 weeks in SEN students' behavior regulations (classroom self-regulation and social skills) using the Child Behavior Rating Scale (CBRS) | 16 weeks
  To increase over 70% of SEN Students' self-regulation and social skills after participated the 16-week SWELE programme.
  The Child Behavior Rating Scale (CBRS) consists of 17 items that measure children's behavioral regulation as illustrated by two subscales: the Classroom Self-Regulation subscale (10 items) and Social Skills subscale (7 items) that assess teachers' perceptions of children's behavioral regulation in social situations.
  Observers/teachers will be asked to rate each item using the following scale (Scale of 1-5; 1 = not at all, 2 = a little, 3 = sometimes, 4= always, 5 = often). The range of score from 17 to 85. Scores The mean of the scale will be calculated with the mean difference will be compared between the baseline and at 16 weeks. The higher score shows a high anxiety level of individual.
Change scores from baseline to 16 weeks in SEN students' playfulness using the Children's Playfulness Scale (CPS) | 16 weeks
  To increase 70% of SEN students' playfulness after participated the 16-week SWELE programme.
  Children's Playfulness Scale (CPS) is a 23-item, and it was used by teachers evaluate the children's behavior. This 5-point Likert scale is designed to assess children's playfulness based on five dimensions: physical spontaneity, social spontaneity, cognitive spontaneity, manifest joy, and sense of humor. Each item poses a statement such as "the child uses unconventional objects in play," which is scored on a 5-point Likert-type scale with responses ranging from "sounds exactly like the child" to "doesn't sound at all like the child".

CONTACTS AND LOCATIONS:
Overall Officials: Regina Lee, PhD, Principal Investigator — Chinese University of Hong Kong

REFERENCES:
- [Background] Lee RLT, Lane S, Brown G, Leung C, Kwok SWH, Chan SWC. Systematic review of the impact of unstructured play interventions to improve young children's physical, social, and emotional wellbeing. Nurs Health Sci. 2020 Jun;22(2):184-196. doi: 10.1111/nhs.12732. PMID 32358875
- [Derived] Lee RLT, Chan SWC, Chong YY, Chau SWH, Choi KC, Chien WT. Effects of a SWELE program for improving mental wellbeing in children and adolescents with special educational needs: protocol of a quasi-experimental study. BMC Pediatr. 2024 Dec 6;24(1):800. doi: 10.1186/s12887-024-05288-8. PMID 39643869